CLINICAL TRIAL: NCT05221567
Title: The Effectiveness of Intensive Psychotherapy for Chronic Depression: A Naturalistic Comparison With Treatment-as-Usual
Brief Title: Intensive Psychotherapy for Chronic Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modum Bad (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ModumBad chronic depression
Record Dates: First submitted 2022-01-21; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Chronic Depression; Persistent Depressive Disorder; Recurrent Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity high dosage inpatient short-term psychodynamic psychotherapy (affect phobia therapy) (Active Comparator): APT and VITA psychotherapy was carried out in accordance with treatment manuals. In addition to weekly individual sessions the inpatient program at both groups contained two 75 min group sessions each week. In addition, VITA had shorter group meetings each morning (15 minutes). Patients in both treatments participated in two physical exercise sessions per week, weekly psycho-educational lectures and art-therapy groups, and both groups finish each week with end of the week status groups. On average, patients in both treatments received seven sessions of therapeutic activity each week. All treatment components, with the exception of the physical exercises, adhered to the APT or VITA treatments, and thus the two intensive treatments were similar in dose but different in content. Medication was managed by psychiatrists, aiming to optimize the psychotropic medication regime, typically by reducing medication use.
  Interventions: Behavioral: Psychotherapy
- Treatment-as-usual (Other): TAU through public services locally, either outpatient treatment from a psychologist/psychiatrist and/or treatment/support from their local general practitioner.
  Interventions: Behavioral: Psychotherapy
- High intensity high dosage inpatient short-term psychodynamic psychotherapy (VITA) (Active Comparator): APT and VITA psychotherapy was carried out in accordance with treatment manuals. In addition to weekly individual sessions the inpatient program at both groups contained two 75 min group sessions each week. In addition, VITA had shorter group meetings each morning (15 minutes). Patients in both treatments participated in two physical exercise sessions per week, weekly psycho-educational lectures and art-therapy groups, and both groups finish each week with end of the week status groups. On average, patients in both treatments received seven sessions of therapeutic activity each week. All treatment components, with the exception of the physical exercises, adhered to the APT or VITA treatments, and thus the two intensive treatments were similar in dose but different in content. Medication was managed by psychiatrists, aiming to optimize the psychotropic medication regime, typically by reducing medication use.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Intensive psychotherapy (i.e., greater number of treatment sessions per time unit)

SUMMARY:
The study evaluates whether Intensive psychotherapy show superior effect on chronic depression over TAU

DETAILED DESCRIPTION:
Background: Accumulating evidence indicates that intensive psychotherapy (i.e., greater number of treatment sessions per time unit) improves outcomes for patients with mental health problems. However, few studies have investigated whether patients with chronic depression (CD) benefit from treatment with higher intensity. The main purpose of this study is to investigate if intensive psychotherapy could improve treatment for patients with chronic depression (CD). The primary research question is whether two intensive psychodynamic inpatient treatments, affect phobia therapy (APT) and VITA, are superior to low intensity treatment (TAU) at completion of treatment. To indicate if a potential difference between intensive treatment and TAU is due to the intensity of the therapy, the study contrasts two therapies with similar intensity, but different theoretical rationales. Methods: 280 patients with CD are included in a naturalistic study. Patients are assessed at four time points; assessment, start of therapy, end of therapy and 1-year follow-up. Three comparisons are performed with patients matched across groups; Intensive treatment (APT + VITA) vs TAU during treatment, APT vs VITA during treatment and APT vs VITA during follow-up. The outcome measure is the BDI-II.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be liberal and similar to clinical practice criteria at the treatment site which includes patients with the characteristics of chronic depression (CD), thus including patients with

* Persistent depressive disorder as defined by the diagnostic and statistical manual of mental disorders (DSM5)
* Recurrent depressive disorder as defined by the International classification of diseases-10 (ICD-10)

Exclusion Criteria:

* Not having utilized reasonably available treatment in proximity to their residence
* A psychotic disorder
* Cluster A or B personality disorder
* Bipolar disorder,
* Ongoing substance abuse,
* Physical brain disorder
* Not having access to TAU while on the 12 week wait-list period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Depressive symptoms | Patients were assessed at four time points; assessment, start of therapy (12 weeks after assessment), end of therapy (24 weeks after assessment) and at 1-year follow-up (76 weeks after assessment).
  Beck depression inventory II (BDI-II) Self-report instrument for assessing severity of depression. 21 items are scored on Likert scale from 0 to 4 (range 0-63). Scores between 14 and 19 indicate mild depression, 20 to 28 indicate moderate depression, and above 29 indicate major depression.

CONTACTS AND LOCATIONS:
Overall Officials: KariAnne Vrabel, PhD, Study Director — Leader Modum Bad Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eielsen M, Ulvenes PG, Rossberg JI, Hostmaelingen A, Soma CS, Wampold BE. The Effectiveness of an Intensive Inpatient Psychotherapy Program for Chronic Depression: A naturalistic comparison with wait list. BMC Psychiatry. 2022 Nov 30;22(1):745. doi: 10.1186/s12888-022-04381-5. PMID 36451114